CLINICAL TRIAL: NCT05488002
Title: The Impact of Pharmacist Counseling and Follow-up on Hypertensive, Diabetic, and Obese Patients in the UAE
Brief Title: Pharmacists Interventions on Patients Diabetic, and Obese Patients in the UAE: Randomized Controlled Trials.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Osama Mohamed Ibrahim, Associate professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC-22-03-17-03
Record Dates: First submitted 2022-06-29; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Hypertension; Diabete Type 2; Obesity; Pharmacist-Patient Relations
Keywords: Hypertension; Diabete Type 2; Pharmacist interventions
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Obesity | interventions — Safety

STUDY DESIGN:
Intervention Model Description: This study comprises 3 trials with the same intervention. Pharmacists will be trained how to recruit patients and perform pharmaceutical interventions. Each pharmacy will be required to recruit 45patients (15 hypertension, 15 diabetes, and 15 obese).
  These patients will be randomized into two groups : intervention, which will receive pharmaceutical intervention and control group, which will receive standard care
  *The general practitioner of each participant will be informed about the study by a letter.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will receive pharmaceutical interventions.
  Hypertensive patients will receive pharmacist recommendations on hypertension Diabetic patients will receive pharmacist recommendations on diabetes Obese patients will receive pharmacist recommendations on obesity
  Interventions: Behavioral: Pharmaceutical intervention
- Control (No Intervention): This arm will receive standard care

INTERVENTIONS:
Behavioral: Pharmaceutical intervention — Pharmacists will provide clinical recommendations to patients allocated to the intervention group. Furthermore, they will monitor patients' parameters and follow-up with them. These interventions include daily medication review, weight, heart monitoring, blood glucose level, follow-up on medication adherence, and even mental status.
  Other Names: Pharmacist recommendations; Heart monitoring; Blood glucose level monitoring; Weight monitoring; Medication adherence follow-up; Coaching on medication use and safety; Coaching on healthy diet; Mental and emotional support
  Arms: Intervention

SUMMARY:
Hypertension, diabetes, and obesity are considered major risk factors for cardiovascular diseases and premature mortality worldwide. Furthermore, they have severe consequences on quality of life among patients. With increasing challenges facing the healthcare systems, pharmacists are well positioned to take on a greater role in the management of chronic diseases.

The present study aims to investigate the impact of pharmacist counselling on the clinical outcomes (weight, mortality, blood pressure, blood glucose) of hypertensive, diabetic, and obese patients.

DETAILED DESCRIPTION:
This will be a multicentric randomized, controlled trial comparing enhanced pharmacist care (which included independent patient assessment, counseling, and follow-up) with usual care in the UAE over a year. Generally, this research project will be conducted on 3 phases;

1. patients who suffer from elevated blood pressure will be Randomised into two groups, of which one of them will receive a standard care and the second one will receive pharmaceutical care. Both will be followed up to 26 weeks (an estimated period to monitor blood pressure change).
2. patients with diabetes will be identified and Randomised using the same approach and followed up to 12 weeks (In order to monitor the HbA1c ).
3. Patients with obesity (BMI is 30 or higher) will be Randomised and followed up to 16 weeks (according to the literature, this is the period required to monitor the BMI change). SPSS V26 will be used for Data analysis.

This research will enable the determination of the effectiveness of pharmacist counseling and follow-up in improving the clinical outcomes of chronic diseases (diabetes, hypertension, and obese) patients, which has never been assessed in the UAE.

* The provided evidence may help in the implementation of a new novel practice in the world, in which the pharmacist's roles are expanded and evolved to include continual counseling on chronic disease patients and follow up. Thus, reducing the burden, and ensure sustainability of the healthcare services in the UAE.
* Publications in peer-reviewed journals (At least 3 papers are expected), both international and local and conference presentations will be attempted to share the findings of our research.

Therefore, the study aims to:

1. To assess the impact of pharmacist counseling on the mortality rate of diabetic, hypertensive and obese patients.
2. To study the impact of pharmacist counseling on the morbidity rate of diabetic, hypertensive and obese patients.
3. To measure the effectiveness of pharmacist counseling on improving the blood pressure of hypertensive patients.
4. To evaluate the benefits of pharmacist counseling on blood glucose level among diabetic patients.
5. To examine the impact of pharmacist recommendations and medication review on the weight and cholesterol level among obese patients.
6. To investigate potential adverse effects may be induced upon pharmacist counseling.
7. To explore any drug-related problems may be induced by pharmacist interventions.
8. To study the satisfaction of diabetic, hypertensive, and obese patients with pharmacist counselling.

ELIGIBILITY:
Inclusion Criteria:

1. age between 45 years and 75 years, BMI: 25 kg ⁄ m2 , treatment with oral hypoglycemic medication for at least 12 months, and a regular visitor of the pharmacy.
2. blood pressure (BP) measurements in the clinic of systolic BP (SBP) <140 mmHg and diastolic BP (DBP) <90 mmHg and they are on established antihypertensive drug treatment for at least 6 months.
3. BMI >30 , seeking to lose weight or improve eating habits will be recruited.

Exclusion Criteria:

1. Younger than 45,, being solely on insulin treatment (no oral hypoglycemic treatment) will also be an exclusion criterion.
2. Pregnancy.
3. breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose | Up to 3 months
  The device used will be glucometer and the results will be expressed in (mmol/L)
Glycosylated haemoglobin (HbA1c) | 12 weeks
  An A1c test result gets reported as a percentage. The number represents the portion of hemoglobin proteins that are glycated, or holding glucose. The higher the percentage, the higher your blood sugar levels have been over the last few months.
  Less than 5.7% means you don't have diabetes. 5.7% to 6.4% signals pre-diabetes. 6.5% or higher means a diabetes diagnosis. 7% or lower is the goal for someone trying to manage their diabetes.
Adherence to oral hypoglycaemic agents | Up to 3 months
  The Medication Adherence Reasons Scale (MAR-Scale) is a 20-item comprehensive scale that was developed to measure medication adherence.
Drug-related problems | Up to 3 months
  We will use a drug-related problems classification system developed by Prof. Salah (AbuRuz, S.M., Bulatova, N.R. & Yousef, A.M. Validation of a comprehensive classification tool for treatment-related problems . Pharm World Sci 28, 222-232 (2006). https://doi.org/10.1007/s11096-006-9048-0
  ) which includes six main categories for treatment-related problems (Indication, Effectiveness, Safety, Knowledge, Adherence and Miscellaneous)
Blood pressure values | Up to 3 months
  Sphygmomanometer will be used to measure systolic and diastolic pressure values.
Weight | 6 months
  It will be reported in Kg
Cholesterol LDL-cholesterol Triglycerides Cholesterol LDL-cholesterol Triglycerides | 6 months
  The cholesterol home test kit will be used and results will be expressed in milligrams (mg) of cholesterol per deciliter (dL) of blood.

SECONDARY OUTCOMES:
Knowledge about diabetes | Up to 3 months
  Diabetes Knowledge Questionnaire (DKQ) will be used
knowledge about hypertension | Up to 3 months
  The HKT is a simple questionnaire for assessing and monitoring HBP knowledge. It is sensitive to differences in blood pressure control status and should provide a valid, reliable, and standardized measure of HBP knowledge with wide relevance.
Medication adherance | Up to 3 months
  he Medication Adherence Reasons Scale (MAR-Scale) is a 20-item comprehensive scale that was developed to measure medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Ibrahim, PhD, Principal Investigator — Associate professor College of Pharmacy Pharmacy Practice & Pharmacotherapeutics

IPD SHARING:
Plan to Share IPD: No